CLINICAL TRIAL: NCT07380841
Title: Comparative Effectiveness of Metformin, Inositol, Dietary Restriction, and Combination Therapy in Polycystic Ovary Syndrome: A 12-Week Prospective Randomized Study
Brief Title: Metformin vs Inositol vs Diet vs Combination Therapy in PCOS
Acronym: PCOS-COMBO (9)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Islamabad Medical and Dental College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCOS-MIDCOMBO-12W-2025; F-1/2015/ERB/SZABMU/1449) (Other: Shaheed Zulfiqar Ali Bhutto Medical University)
Record Dates: First submitted 2026-01-24; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Polycystic Ovary Syndrome; Insulin Resistance; Metabolic Syndrome
Keywords: PCOS, Metformin, Myo-inositol, Dietary Restriction, Insulin Resistance, Weight Loss, Combination Therapy
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance; Metabolic Syndrome; Weight Loss | interventions — Metformin; Inositol; Diet Therapy; Caloric Restriction; Diet, Reducing

STUDY DESIGN:
Intervention Model Description: Four-arm, randomized, parallel-group comparative trial.
Masking Description: Due to the nature of the interventions (drug and lifestyle), the study was conducted in an open-label manner.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Metformin Group (Experimental): Participants will receive metformin hydrochloride tablets, 500 mg orally twice daily (total daily dose 1000 mg) after meals for 12 weeks. This arm evaluates the effect of metformin monotherapy on metabolic, hormonal, and clinical outcomes in women with polycystic ovary syndrome (PCOS).
  Interventions: Drug: Metformin Hydrochloride
- Inositol Group (Experimental): Participants will receive myo-inositol powder/sachets, 2 g orally twice daily (total daily dose 4 g) for 12 weeks. This arm evaluates the effect of inositol monotherapy on insulin resistance, hormonal profile, and clinical features of PCOS.
  Interventions: Dietary Supplement: Myo-Inositol
- Dietary Restriction Group (Experimental): Participants will follow a structured calorie-restricted diet (approximately 1200-1500 kcal/day, individualized according to baseline BMI), designed and supervised by the study team, for 12 weeks. No pharmacological treatment will be given. This arm evaluates the effect of dietary intervention alone on anthropometric, metabolic, and reproductive outcomes in PCOS.
  Interventions: Behavioral: Dietary Restriction
- Combination Therapy Group (Experimental): Participants will receive metformin hydrochloride tablets 500 mg orally twice daily plus myo-inositol 2 g orally twice daily, along with the same structured calorie-restricted diet (1200-1500 kcal/day) for 12 weeks. This arm evaluates the combined effect of pharmacological and lifestyle intervention on metabolic, hormonal, and clinical outcomes in PCOS.
  Interventions: Combination Product: Metformin + Myo-inositol + Dietary Restriction

INTERVENTIONS:
Drug: Metformin Hydrochloride — Metformin is an insulin-sensitizing biguanide used to improve glucose metabolism and reduce insulin resistance in women with polycystic ovary syndrome. It is administered orally as part of the study protocol to evaluate its effects on metabolic, hormonal, and reproductive outcomes.
  Other Names: Glucophage
  Arms: Metformin Group
Dietary Supplement: Myo-Inositol — Myo-inositol is a nutritional supplement involved in insulin signaling pathways and ovarian function. It is used in this study to assess its effect on insulin sensitivity, hormonal profile, and clinical features of polycystic ovary syndrome.
  Other Names: Inositol; Vitamin B8
  Arms: Inositol Group
Behavioral: Dietary Restriction — A structured, supervised calorie-restricted dietary program is used as a lifestyle intervention to improve weight, metabolic parameters, and reproductive function in women with polycystic ovary syndrome.
  Other Names: Calorie-restricted diet; Weight Reduction Diet
  Arms: Dietary Restriction Group
Combination Product: Metformin + Myo-inositol + Dietary Restriction — This intervention combines pharmacological insulin sensitization and nutritional supplementation with lifestyle modification to evaluate the synergistic effect on metabolic, hormonal, and clinical outcomes in women with polycystic ovary syndrome.
  Other Names: Combined lifestyle and pharmacological intervention
  Arms: Combination Therapy Group

SUMMARY:
Polycystic ovary syndrome (PCOS) is a common condition that can cause irregular periods, excess male-type hormones, weight gain, and insulin resistance. This study will compare four commonly used approaches for PCOS management: metformin, inositol, a calorie-restricted diet, and a combination of all three.

A total of 192 women aged 18-35 years with PCOS (diagnosed using Rotterdam criteria) will be randomly assigned to one of four groups for 12 weeks: (A) metformin, (B) myo-inositol plus D-chiro-inositol, (C) calorie-restricted diet, or (D) combination therapy (metformin + inositol + diet). The study will assess changes in body weight, body mass index (BMI), waist circumference, fasting glucose, fasting insulin, insulin resistance (HOMA-IR), and menstrual regularity. Hormonal measures and safety outcomes will also be evaluated. The goal is to determine which approach provides the greatest overall metabolic and reproductive benefit in women with PCOS.

DETAILED DESCRIPTION:
This is a 12-week, prospective, randomized, parallel-group controlled clinical trial conducted at an academic tertiary-care center in Islamabad, Pakistan (July-October 2025). The trial compares the independent and combined effects of metformin, inositol, and calorie restriction on metabolic, anthropometric, hormonal, and reproductive outcomes in women with polycystic ovary syndrome (PCOS).

Participants A total of 192 reproductive-aged women (18-35 years) with PCOS diagnosed by Rotterdam criteria (≥2 of: oligo/anovulation, clinical/biochemical hyperandrogenism, polycystic ovarian morphology on ultrasound) will be enrolled. Key exclusions include thyroid dysfunction, hyperprolactinemia, congenital adrenal hyperplasia, Cushing syndrome, hepatic/renal impairment, pregnancy or lactation, and use of hormonal therapy or insulin-sensitizing agents within the preceding 3 months.

Randomization and masking Participants will be randomized in a 1:1:1:1 allocation (n=48 per group) using a computer-generated sequence, with allocation concealment using sequentially numbered, opaque, sealed envelopes. Due to the nature of interventions, participant blinding is not feasible; however, laboratory personnel and data analysts will remain blinded to group assignment.

Interventions (12 weeks) Group A (Metformin): metformin 1500-2000 mg/day orally, titrated according to gastrointestinal tolerance.

Group B (Inositol): myo-inositol 2 g plus D-chiro-inositol 50 mg, taken twice daily.

Group C (Calorie-restricted diet): individualized dietary counseling targeting 1200-1500 kcal/day with emphasis on low-glycemic carbohydrates, lean protein, and high-fiber foods.

Group D (Combination): metformin + inositol + calorie-restricted diet as above. Participants will be followed every two weeks for adherence assessment and adverse event monitoring. Medication adherence will be assessed by pill counts. Dietary adherence will be assessed using weekly dietary logs and summarized as percent compliance with prescribed caloric intake.

Outcomes

Primary outcomes assessed at baseline and 12 weeks include:

Anthropometric measures: weight, BMI, waist circumference; Metabolic measures: fasting glucose, fasting insulin, and insulin resistance (HOMA-IR; calculated as [fasting insulin × fasting glucose]/405); Menstrual regularity, defined as cycle length 21-35 days during the final four weeks of the intervention.

Secondary outcomes include serum total testosterone, LH, FSH, LH/FSH ratio, Ferriman-Gallwey score, adherence, and adverse events. Fasting blood samples will be collected and hormonal assays performed using standardized chemiluminescence immunoassay platforms.

Statistical approach Normality will be assessed using Shapiro-Wilk tests. Continuous variables will be summarized as mean ± SD. Within-group changes will be analyzed using paired t-tests. Between-group comparisons will use one-way ANOVA with Tukey HSD post-hoc testing. Effect sizes will be reported as partial eta-squared (η²). Categorical outcomes (e.g., menstrual regularity) will be compared using chi-square tests. Statistical significance will be defined as p < 0.05. Analyses will follow CONSORT reporting principle

ELIGIBILITY:
Inclusion Criteria:Females aged 18 to 40 years. Diagnosed with polycystic ovary syndrome (PCOS) based on Rotterdam criteria (at least two of the following: oligo/anovulation, hyperandrogenism, polycystic ovaries on ultrasound).

Body mass index (BMI) ≥ 18.5 kg/m². Willing to participate and provide written informed consent. Willing to comply with study procedures and follow-up visits.

-

Exclusion Criteria:

Pregnancy or lactation. Known diabetes mellitus, thyroid disease, hyperprolactinemia, Cushing's syndrome, or other endocrine disorders.

Use of metformin, inositol, hormonal therapy, or weight-loss drugs within the last 3 months.

History of renal, hepatic, or cardiovascular disease. Known hypersensitivity to metformin or inositol. Participation in another clinical trial within the last 3 months. Any serious medical or psychiatric condition that, in the investigator's opinion, would interfere with study participation.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only women diagnosed with polycystic ovary syndrome (PCOS) according to standard diagnostic criteria are eligible for participation in this study
Enrollment: 192 (Actual)
Dates: Start 2025-05-21 (Actual); Primary Completion 2025-11-11 (Actual); Study Completion 2026-01-13 (Actual)

PRIMARY OUTCOMES:
Change in insulin resistance (HOMA-IR) | Baseline to 12 weeks
  Mean change in insulin resistance as measured by the Homeostatic Model Assessment of Insulin Resistance (HOMA-IR), calculated from fasting plasma glucose and fasting serum insulin levels, comparing baseline values to 12-week follow-up among the four treatment groups (metformin, inositol, dietary restriction, and combination therapy).

SECONDARY OUTCOMES:
Change in body weight and body mass index (BMI) | Baseline to 12 weeks
  Mean change in body weight (kg) and body mass index (kg/m²) from baseline to 12 weeks.
Change in menstrual cycle regularity | Baseline to 12 weeks
  Proportion of participants achieving regular menstrual cycles or improvement in cycle regularity over the 12-week intervention period.Baseline to 12 weeks
Change in serum androgen levels | Baseline to 12 weeks
  Mean change in serum total testosterone levels from baseline to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shemaila Saleem, Study Director — Shaheed Zulfiqar Ali Bhutto Medical University
Locations (1):
- Pakistan Institute of Health Sciences / Islamabad Medical and Dental College (IMDC), Islamabad, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the results reported in this study, including demographic, clinical, biochemical, and outcome variables, will be made available to qualified researchers upon reasonable request. Data will be shared in a de-identified format to protect participant confidentiality. Requests will be reviewed by the principal investigator and the institutional ethics committee.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The data will be available beginning 6 months after publication of the primary results and will remain available for 5 years thereafter.
Access Criteria: Access to the data will be granted to researchers who provide a methodologically sound proposal, obtain approval from the principal investigator and the institutional ethics committee, and sign a data use agreement. Data will be used only for non-commercial, academic research purposes.